CLINICAL TRIAL: NCT00928083
Title: A Phase I Study To Investigate The Safety, Tolerability And Pharmacokinetic Profile Of OZ439 In Healthy Male and Female Subjects
Brief Title: A Study to Investigate the Safety, Tolerability and Pharmacokinetics of OZ439 in Healthy Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MMV_OZ439_09_001
Record Dates: First submitted 2009-06-24; First posted 2009-06-25 (Estimated); Results first posted 2015-01-08 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Malaria Falciparum; Malaria Vivax; Healthy Volunteers
Keywords: Phase I; Safety and tolerability; Pharmacokinetic; synthetic peroxide; trioxolane; treatment of erythrocytic stages of malaria
MeSH Terms: conditions — Malaria, Falciparum; Malaria, Vivax | interventions — artefenomel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (17):
- Part A - 50 mg Single Dose (Experimental): OZ439 Single doses of 50mg (capsules)
  Interventions: Drug: OZ439 50mg API capsules
- Part A - 100mg Single Dose (Experimental): OZ439 Single doses of 100mg (capsules)
  Interventions: Drug: OZ439 100mg API capsules
- Part A - 200mg Single Dose (Experimental): OZ439 Single doses of 200mg (capsules)
  Interventions: Drug: OZ439 200mg API capsules
- Part A - 400mg Single Dose (Experimental): OZ439 Single doses of 400mg (capsules)
  Interventions: Drug: OZ439 400mg API capsules
- Part A - 400mg Single Dose + Food (Experimental): OZ439 Single doses of 400mg (capsules) administered with food.
  Interventions: Drug: OZ439 400mg API capsules
- Part A - 400mg AD Single Dose (Experimental): OZ439 Single doses of 400mg (aqueous dispersion)
  Interventions: Drug: OZ439 400mg aqueous dispersion
- Part A - 800mg Single Dose (Experimental): OZ439 Single doses of 800mg (capsules)
  Interventions: Drug: OZ439 800mg API capsules
- Part A - 800mg AD Single Dose (Experimental): OZ439 Single doses of 800mg (aqueous dispersion)
  Interventions: Drug: OZ439 800mg aqueous dispersion
- Part A - 1200mg Single Dose (Experimental): OZ439 Single doses of 1200mg (capsules)
  Interventions: Drug: OZ439 1200mg API capsules
- Part A - 1600mg AD Single Dose (Experimental): OZ439 Single doses of 800mg (aqueous dispersion)
  Interventions: Drug: OZ439 1600mg aqueous dispersion
- Part A - Placebo (Placebo Comparator): Placebo control for Single rising Part A
  Interventions: Drug: Placebo
- Part B - 800mg AD Single Dose Fed (Experimental): Single dose of OZ439 800mg aqueous dispersion administered under fed conditions
  Interventions: Drug: OZ439 800mg aqueous dispersion
- Part B - 800mg AD Single Dose Fast (Experimental): Single dose of OZ439 800mg aqueous dispersion administered under fast conditions
  Interventions: Drug: OZ439 800mg aqueous dispersion
- Part C - 200mg AD Multiple Dose (Experimental): 200mg aqueous solution OZ439 or placebo once daily for 3 days fasted
  Interventions: Drug: OZ439 200mg aqueous dispersion
- Part C - 400mg AD Multiple Dose (Experimental): 400mg aqueous solution OZ439 or placebo once daily for 3 days fasted
  Interventions: Drug: OZ439 400mg aqueous dispersion
- Part C - 800mg AD Multiple Dose (Experimental): 800mg aqueous solution OZ439 or placebo once daily for 3 days fasted
  Interventions: Drug: OZ439 800mg aqueous dispersion
- Part C - Placebo (Placebo Comparator): Placebo control for Multiple rising Part C
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OZ439 50mg API capsules
  Other Names: OZ439
  Arms: Part A - 50 mg Single Dose
Drug: OZ439 200mg API capsules
  Other Names: OZ439
  Arms: Part A - 200mg Single Dose
Drug: OZ439 400mg aqueous dispersion
  Arms: Part A - 400mg AD Single Dose; Part C - 400mg AD Multiple Dose
Drug: OZ439 800mg aqueous dispersion
  Other Names: OZ439
  Arms: Part A - 800mg AD Single Dose; Part B - 800mg AD Single Dose Fast; Part B - 800mg AD Single Dose Fed; Part C - 800mg AD Multiple Dose
Drug: OZ439 100mg API capsules — OZ439 100mg (2x50mg API capsules)
  Other Names: OZ439
  Arms: Part A - 100mg Single Dose
Drug: OZ439 400mg API capsules — OZ439 400mg (2x200mg API capsules)
  Other Names: OZ439
  Arms: Part A - 400mg Single Dose; Part A - 400mg Single Dose + Food
Drug: OZ439 1600mg aqueous dispersion
  Other Names: OZ439
  Arms: Part A - 1600mg AD Single Dose
Drug: OZ439 800mg API capsules — OZ439 800mg (4x200 API capsules)
  Other Names: OZ439
  Arms: Part A - 800mg Single Dose
Drug: OZ439 1200mg API capsules — OZ439 1200mg (6x200mg API capsules)
  Other Names: OZ439
  Arms: Part A - 1200mg Single Dose
Drug: Placebo
  Arms: Part A - Placebo; Part C - Placebo
Drug: OZ439 200mg aqueous dispersion
  Other Names: OZ439
  Arms: Part C - 200mg AD Multiple Dose

SUMMARY:
OZ439 is a synthetic trioxolane that has potential value as a peroxide antimalarial agent.

This was a Phase I, single-centre, multi-component, double-blind, randomised, placebo-controlled study in healthy male and female subjects. The study was conducted in 3 parts:

* Part A investigated the safety, tolerability and pharmacokinetics (PK) of single oral escalating doses of OZ439. Up to 6 dose levels will be investigated to estimate dose proportionality.
* Part B, the effect of food on a single oral dose of OZ439 was investigated in a 2-way crossover design.
* Part C investigated the safety, tolerability and PK profile of multiple oral doses of OZ439.

The starting oral dose was 50 mg and the maximum single dose to be administered did not exceed 1600 mg per subject. The maximum duration of dosing proposed was 3 days.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male//female subjects between 18- 55 years of age (inclusive).
2. Body mass Index (BMI) between 18 - 30 kg/m2, inclusive; and a total body weight >60 kg (132 lbs).
3. Healthy as determined by pre-study medical history, PE, 12 Lead ECG.
4. Females of childbearing potential must use 1 of birth control methods throughout study and for 30 days after last dose of study drug:

   1. Surgically sterile (bilateral tubal ligation, hysterectomy, bilateral oophorectomy) 6 months minimum prior to first dose of study drug.
   2. Intrauterine device (IUD) in place for at least 3 months prior to first dose of study drug.
   3. Barrier methods (condom or diaphragm) with spermicide starting at least 14 days prior to first dose of study drug through 30 days after last dose of study drug.
   4. Surgical sterilization of the partner(s) (vasectomy with zero sperm count for 6 months minimum prior to the first dose of study drug).
   5. Hormonal contraceptives starting at least 3 months prior to first dose of study drug. In addition, subjects must agree to use a barrier method (condom or diaphragm) with spermicide at least 14 days prior to first dose of study drug through 30 days after the last dose of study drug.
5. Post-menopausal women with amenorrhea for at least 1 year will be eligible confirmed by FSH.
6. Male subjects must agree to use double barrier method of contraception, from time of first dose of study drug through 90 days after last dose of study drug and must also agree to not donate sperm for 90 days after last dose of study drug. Clinical laboratory tests within the reference ranges.
7. Able/willing to give written informed consent.
8. Willing/to adhere to lifestyle guideline restrictions outlined in protocol.
9. Willing and able to be confined to Clinical Research Unit as required by the protocol.

Exclusion Criteria:

1. Evidence/history of clinically significant oncologic, pulmonary, hepatic, cardiovascular, hematologic, metabolic, neurological, immunologic, nephrologic, endocrine, psychiatric disease, current infection.
2. Evidence/history of clinically significant gastrointestinal (some exclusions exist) disease, current infection.
3. Any condition that affecting drug absorption, e.g., gastrectomy.
4. History of post-antibiotic colitis.
5. Breast feeding.
6. QTc greater than 450 msec for males and 470 msec for females as corrected by the Bazett formula.
7. History of drug or alcohol abuse within the past 2 years prior to Screening.
8. Tobacco users
9. Received investigational drug/ participated in another research study within 30 days of first dose of study drug in any part of study.
10. Use of prescription drugs within 14 days prior to the first dose of study drug in Period 1, or need for any antibiotic during study.
11. Received any non prescription meds, vitamins, herbal/dietary supplements within 7 days of administration of first dose of study drug in Period 1 (exceptions exist)
12. Consumed alcohol within 72 hours of Day -1 in any part of study, or have a positive alcohol screen at screening or each admission to Clinical Research Unit (CRU).
13. Consumed grapefruit juice or juices containing grapefruit or ate grapefruit within 7 days prior to first dose of study drug in any part of study.
14. Positive serum pregnancy test at the Screening Visit or on Day -1 prior to inclusion in any part of the study.
15. Positive test for HIV-1, HBsAg,HCV.
16. Positive urine drug screen at Screening or admission to CRU.
17. History of intolerance/ hypersensitivity to artemisinins.
18. Likelihood of requiring treatment during study period with drugs not permitted by protocol.
19. Subjects who have donated blood or experienced significant blood loss within 60 days of screening for study.
20. Subjects whose hemoglobin is <12.5 g/dL for males/ <11.5 g/dL for females.
21. Any concern by investigator regarding safe participation of the subject in study or for any other reason investigator considers subject inappropriate for participation in study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2009-04; Primary Completion 2009-10 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Moehrle, PhD, Study Director — Medicines for Malaria Venture; Maria Gutierrez, MD, Principal Investigator — Comprehensive Phase One Miramar, 3400 Enterprise Way, Miramar, FL 33025
Locations (1):
- Comprehensive Phase One Miramar; 3400 Enterprise Way, Miramar, Florida, United States

REFERENCES:
- [Result] Moehrle JJ, Duparc S, Siethoff C, van Giersbergen PL, Craft JC, Arbe-Barnes S, Charman SA, Gutierrez M, Wittlin S, Vennerstrom JL. First-in-man safety and pharmacokinetics of synthetic ozonide OZ439 demonstrates an improved exposure profile relative to other peroxide antimalarials. Br J Clin Pharmacol. 2013 Feb;75(2):524-37. doi: 10.1111/j.1365-2125.2012.04368.x. PMID 22759078

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A - OZ439 Single Dose - Cohort 1: OZ439 50 mg then 200 mg, then 800 mg, then 1600 mg, then Placebo
- Part A - OZ439 Single Dose - Cohort 2: OZ439 50 mg, then 100 mg, then 400 mg, then 1200 mg, then Placebo
- Part A - OZ439 Single Dose - Cohort 3: Oral Dispersion OZ439 50-1600 mg
- Part B - Food Effect - Cohort 1: Food Effect - Cohort 1 800mg OZ439 Fasted then Fed
- Part B - Food Effect - Cohort 2: Food Effect - Cohort 2 800mg OZ439 Fed then Fasted
- Part C - 200mg OZ439 Multiple Dose: 200mg OZ439 for 3 consecutive days
- Part C - 400mg OZ439 Multiple Dose: OZ439 400mg for 3 consecutive days
- Part C - 800mg OZ439 Multiple Dose: OZ439 800mg for 3 consecutive days
- Part C - Placebo: Part C - Placebo
Period: Overall Study
Arm/Group | Part A - OZ439 Single Dose - Cohort 1 | Part A - OZ439 Single Dose - Cohort 2 | Part A - OZ439 Single Dose - Cohort 3 | Part B - Food Effect - Cohort 1 | Part B - Food Effect - Cohort 2 | Part C - 200mg OZ439 Multiple Dose | Part C - 400mg OZ439 Multiple Dose | Part C - 800mg OZ439 Multiple Dose | Part C - Placebo
Started | 10 | 8 | 8 | 6 | 7 | 6 | 6 | 6 | 6
Completed | 6 | 8 | 8 | 5 | 6 | 6 | 6 | 6 | 6
Not Completed | 4 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part A - OZ439 Single Rising Dose: Included 3 Cohorts, where subjects in cohorts 1 and 2 were randomized to a treatment sequence, receiving doses of OZ439 on four occasions and placebo on one occasion, and subjects in Cohort 3 were administered increasing doses of the oral dispersion.
- Part B - OZ439 Food Effect: Subjects were randomized to sequence groups, "fasted/fed or fed/fasted" while receiving a single dose of 800 mg OZ439.
- Part C - OZ439 Multiple Rising Dose: Subjects were assigned to individual dose cohorts (200, 400 and 800 mg OZ439) and placebo.
- Total: Total of all reporting groups
Arm/Group | Part A - OZ439 Single Rising Dose | Part B - OZ439 Food Effect | Part C - OZ439 Multiple Rising Dose | Total
Number analyzed (Participants) | 26 | 13 | 24 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.6 (10.35) | 33.7 (8.49) | 40.1 (10.17) | 36.5 (9.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 9 | 23
  Male | 21 | 4 | 15 | 40
Region of Enrollment [Number; unit: participants]
  United States | 26 | 13 | 24 | 63

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Safety/Tolerability evaluation took into account the recorded AE profile, clinical laboratory safety tests, vital signs, 12 lead and continuous (Parts A and C) ECG monitoring, audiometry/Brainstem Auditory Evoked Potentials (BAEP) parameters (Parts A and C) including any additional tests required to evaluate any safety concerns.
Time Frame: From screening and at 10 (+/-2) days after last dose of study medication
Measure: Number; unit: participants
Groups:
- Part A - 50 mg Single Dose: OZ439 Single doses of 50mg (capsules)
  OZ439 50mg API capsules
- Part A - 200mg Single Dose: OZ439 Single doses of 200mg (capsules)
  OZ439 200mg API capsules
- Part A - 400mg AD Single Dose: OZ439 Single doses of 400mg (aqueous dispersion)
  OZ439 400mg aqueous dispersion
- Part A - 800mg AD Single Dose: OZ439 Single doses of 800mg (aqueous dispersion)
  OZ439 800mg aqueous dispersion
- Part A - 1600mg AD Single Dose: OZ439 Single doses of 800mg (aqueous dispersion)
  OZ439 1600mg aqueous dispersion
- Part A - Placebo: Placebo control for Single rising Part A
  Placebo
- Part B - 800mg AD Single Dose Fed: Single dose of OZ439 800mg aqueous dispersion administered under fed conditions
  OZ439 800mg aqueous dispersion
- Part B - 800mg AD Single Dose Fast: Single dose of OZ439 800mg aqueous dispersion administered under fast conditions
  OZ439 800mg aqueous dispersion
- Part C - 200mg AD Multiple Dose: 200mg aqueous solution OZ439 or placebo once daily for 3 days fasted
  OZ439 200mg aqueous dispersion
- Part C - 400mg AD Multiple Dose: 400mg aqueous solution OZ439 or placebo once daily for 3 days fasted
  OZ439 400mg aqueous dispersion
- Part C - 800mg AD Multiple Dose: 800mg aqueous solution OZ439 or placebo once daily for 3 days fasted
  OZ439 800mg aqueous dispersion
- Part C - Placebo: Placebo control for Multiple rising Part C
  Placebo
Arm/Group | Part A - 50 mg Single Dose | Part A - 100mg Single Dose | Part A - 200mg Single Dose | Part A - 400mg Single Dose | Part A - 400mg Single Dose + Food | Part A - 400mg AD Single Dose | Part A - 800mg Single Dose | Part A - 800mg AD Single Dose | Part A - 1200mg Single Dose | Part A - 1600mg AD Single Dose | Part A - Placebo | Part B - 800mg AD Single Dose Fed | Part B - 800mg AD Single Dose Fast | Part C - 200mg AD Multiple Dose | Part C - 400mg AD Multiple Dose | Part C - 800mg AD Multiple Dose | Part C - Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 7 | 6 | 5 | 8 | 6 | 6 | 6 | 17 | 12 | 12 | 6 | 6 | 6 | 6
participants | 1 | 0 | 2 | 0 | 0 | 1 | 2 | 1 | 1 | 5 | 4 | 3 | 4 | 3 | 1 | 4 | 0

2. Secondary Outcome: OZ439 AUC0-t
Description: Area under the plasma concentration-time curve from zero to time t of the last measured concentration above the limit of quantification (AUC0-t).
Time Frame: Samples collected from Pre-dose up to 96h post dose
Population: Pharmacokinetics Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.h/ml
Arm/Group | Part A - 50 mg Single Dose | Part A - 100mg Single Dose | Part A - 200mg Single Dose | Part A - 400mg Single Dose | Part A - 400mg AD Single Dose | Part A - 800mg Single Dose | Part A - 800mg AD Single Dose | Part A - 1200mg Single Dose | Part A - 1600mg AD Single Dose | Part B - 800mg AD Single Dose Fed | Part B - 800mg AD Single Dose Fast | Part C - 200mg AD Multiple Dose | Part C - 400mg AD Multiple Dose | Part C - 800mg AD Multiple Dose
Number analyzed (Participants) | 8 | 8 | 8 | 7 | 5 | 8 | 6 | 6 | 6 | 12 | 12 | 6 | 6 | 6
ng.h/ml | 102 (133.7) | 249 (145.4) | 890 (89.1) | 1130 (186.6) | 5430 (72) | 3010 (115.7) | 9630 (56.9) | 6530 (172.4) | 17500 (70.1) | 23100 (48.9) | 7590 (64.7) | 3060 (60.1) | 7990 (57.5) | 13700 (46.0)

3. Secondary Outcome: OZ439 AUC0-∝
Description: Area under the plasma concentration-time curve from zero to infinity (AUC0-∝).
Time Frame: Samples collected from Pre-dose up to 96h post dose
Population: Pharmacokinetics Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.h/ml
Arm/Group | Part A - 50 mg Single Dose | Part A - 100mg Single Dose | Part A - 200mg Single Dose | Part A - 400mg Single Dose | Part A - 400mg AD Single Dose | Part A - 800mg Single Dose | Part A - 800mg AD Single Dose | Part A - 1200mg Single Dose | Part A - 1600mg AD Single Dose | Part B - 800mg AD Single Dose Fed | Part B - 800mg AD Single Dose Fast | Part C - 200mg AD Multiple Dose | Part C - 400mg AD Multiple Dose | Part C - 800mg AD Multiple Dose
Number analyzed (Participants) | 8 | 8 | 8 | 7 | 5 | 8 | 6 | 6 | 6 | 12 | 12 | 6 | 6 | 6
ng.h/ml | NA (NA) — Insufficient data points for calculation | NA (NA) — Insufficient data points for calculation | NA (NA) — Insufficient data points for calculation | NA (NA) — Insufficient data points for calculation | 5540 (71.3) | 4690 (43.5) | 9790 (56.7) | 9130 (136.8) | 18400 (68) | 23900 (49) | 8080 (68.7) | NA (NA) — Insufficient data points for calculation | NA (NA) — Insufficient data points for calculation | NA (NA) — Insufficient data points for calculation

4. Secondary Outcome: OZ439 Cmax
Description: Maximum observed plasma drug concentration (Cmax).
Time Frame: Samples collected from Pre-dose up to 96h post dose
Population: Pharmacokinetics Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | Part A - 50 mg Single Dose | Part A - 100mg Single Dose | Part A - 200mg Single Dose | Part A - 400mg Single Dose | Part A - 400mg AD Single Dose | Part A - 800mg Single Dose | Part A - 800mg AD Single Dose | Part A - 1200mg Single Dose | Part A - 1600mg AD Single Dose | Part B - 800mg AD Single Dose Fed | Part B - 800mg AD Single Dose Fast | Part C - 200mg AD Multiple Dose | Part C - 400mg AD Multiple Dose | Part C - 800mg AD Multiple Dose
Number analyzed (Participants) | 8 | 8 | 8 | 7 | 5 | 8 | 6 | 6 | 6 | 12 | 12 | 6 | 6 | 6
ng/ml | 17.4 (84.7) | 34.2 (173.5) | 102 (82.9) | 135 (164.9) | 566 (53.9) | 315 (121.8) | 917 (35.6) | 701 (154.7) | 1340 (44.5) | 2220 (52.6) | 730 (61.1) | 342 (52.5) | 764 (46.6) | 1390 (51.7)

5. Secondary Outcome: OZ439 Tmax
Description: Time to maximum observed plasma drug concentration of OZ439
Time Frame: Samples collected from Pre-dose up to 96h post dose
Population: Pharmacokinetics Population
Measure: Median (Full Range); unit: hours
Arm/Group | Part A - 50 mg Single Dose | Part A - 100mg Single Dose | Part A - 200mg Single Dose | Part A - 400mg Single Dose | Part A - 400mg AD Single Dose | Part A - 800mg Single Dose | Part A - 800mg AD Single Dose | Part A - 1200mg Single Dose | Part A - 1600mg AD Single Dose | Part B - 800mg AD Single Dose Fed | Part B - 800mg AD Single Dose Fast | Part C - 200mg AD Multiple Dose | Part C - 400mg AD Multiple Dose | Part C - 800mg AD Multiple Dose
Number analyzed (Participants) | 8 | 8 | 8 | 7 | 5 | 8 | 6 | 6 | 6 | 12 | 12 | 6 | 6 | 6
hours | 3 [2 to 6] | 5 [3 to 12] | 3.5 [3 to 6] | 3 [2 to 6] | 3 [2 to 4] | 3 [2 to 4] | 3 [3 to 6] | 3 [2 to 6] | 5 [2 to 6] | 5 [2 to 7] | 3 [2 to 5] | 3 [2 to 5] | 3 [2 to 5] | 3 [2 to 5]

6. Secondary Outcome: OZ439 t1/2
Description: Apparent terminal half-life (t1/2)
Time Frame: Samples collected from Pre-dose up to 96h post dose
Population: Pharmacokinetics Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part A - 50 mg Single Dose | Part A - 100mg Single Dose | Part A - 200mg Single Dose | Part A - 400mg Single Dose | Part A - 400mg AD Single Dose | Part A - 800mg Single Dose | Part A - 800mg AD Single Dose | Part A - 1200mg Single Dose | Part A - 1600mg AD Single Dose | Part B - 800mg AD Single Dose Fed | Part B - 800mg AD Single Dose Fast | Part C - 200mg AD Multiple Dose | Part C - 400mg AD Multiple Dose | Part C - 800mg AD Multiple Dose
Number analyzed (Participants) | 8 | 8 | 8 | 7 | 5 | 8 | 6 | 6 | 6 | 12 | 12 | 6 | 6 | 6
hours | NA (NA) — Below level of detection | NA (NA) — Below level of detection | NA (NA) — Below level of detection | NA (NA) — Below level of detection | 31.2 (33.5) | 27.9 (24.1) | 25.2 (25.8) | 31.6 (46.9) | 30.7 (41.9) | 31.7 (30.1) | 38.8 (50.2) | 41.7 (18.2) | 40.8 (31.4) | 37.8 (28.6)

7. Secondary Outcome: OZ439 Rac
Description: Accumulation index is the ratio of drug exposure observed during a dosing interval at steady-state divided by drug exposure after a single first dose, as described by the following equations:
  Accumulation index (Rac) = AUC0-(Day 3)/ AUC0-(Day 1)
Time Frame: Samples collected from Pre-dose up to 96h post dose
Population: Pharmacokinetics Population received multiple dosing only. This PK parameter is not applicable in a single dose setting.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Part C - 200mg AD Multiple Dose | Part C - 400mg AD Multiple Dose | Part C - 800mg AD Multiple Dose
Number analyzed (Participants) | 6 | 6 | 6
ratio | 1.16 (18.7) | 1.76 (29.9) | 1.43 (26.0)

ADVERSE EVENTS:
Time Frame: Adverse event monitoring throughout the admission period.
Arm/Group | Part A - 50 mg Single Dose | Part A - 100mg Single Dose | Part A - 200mg Single Dose | Part A - 400mg Single Dose | Part A - 400mg Single Dose + Food | Part A - 400mg AD Single Dose | Part A - 800mg Single Dose | Part A - 800mg AD Single Dose | Part A - 1200mg Single Dose | Part A - 1600mg AD Single Dose | Part A - Placebo | Part B - 800mg AD Single Dose Fed | Part B - 800mg AD Single Dose Fast | Part C - 200mg AD Multiple Dose | Part C - 400mg AD Multiple Dose | Part C - 800mg AD Multiple Dose | Part C - Placebo
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/7 | 0/6 | 0/5 | 0/8 | 0/6 | 0/6 | 0/6 | 1/17 | 0/12 | 0/12 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 1/8 | 0/8 | 2/8 | 0/7 | 0/6 | 1/5 | 2/8 | 1/6 | 1/6 | 5/6 | 4/17 | 3/12 | 4/12 | 3/6 | 1/6 | 4/6 | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A - 50 mg Single Dose (N=8) | Part A - 100mg Single Dose (N=8) | Part A - 200mg Single Dose (N=8) | Part A - 400mg Single Dose (N=7) | Part A - 400mg Single Dose + Food (N=6) | Part A - 400mg AD Single Dose (N=5) | Part A - 800mg Single Dose (N=8) | Part A - 800mg AD Single Dose (N=6) | Part A - 1200mg Single Dose (N=6) | Part A - 1600mg AD Single Dose (N=6) | Part A - Placebo (N=17) | Part B - 800mg AD Single Dose Fed (N=12) | Part B - 800mg AD Single Dose Fast (N=12) | Part C - 200mg AD Multiple Dose (N=6) | Part C - 400mg AD Multiple Dose (N=6) | Part C - 800mg AD Multiple Dose (N=6) | Part C - Placebo (N=6)
Influenza (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A - 50 mg Single Dose (N=8) | Part A - 100mg Single Dose (N=8) | Part A - 200mg Single Dose (N=8) | Part A - 400mg Single Dose (N=7) | Part A - 400mg Single Dose + Food (N=6) | Part A - 400mg AD Single Dose (N=5) | Part A - 800mg Single Dose (N=8) | Part A - 800mg AD Single Dose (N=6) | Part A - 1200mg Single Dose (N=6) | Part A - 1600mg AD Single Dose (N=6) | Part A - Placebo (N=17) | Part B - 800mg AD Single Dose Fed (N=12) | Part B - 800mg AD Single Dose Fast (N=12) | Part C - 200mg AD Multiple Dose (N=6) | Part C - 400mg AD Multiple Dose (N=6) | Part C - 800mg AD Multiple Dose (N=6) | Part C - Placebo (N=6)
Atrioventricular Block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Disconfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal Hypermotility (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat Irritation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral Herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Creatine Phosphokinase Increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Pressure Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic Pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Syncope Vasovagal (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less